CLINICAL TRIAL: NCT07185854
Title: Acupuncture Combined With Artificial Tears Compared With Artificial Tears Alone in Moderate Dry Eye: A Randomized Controlled Trial
Brief Title: Medical vs Acupuncture for Dry Eye
Acronym: ADET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nadide Koca (Other)
Responsible Party: Sponsor-Investigator, Nadide Koca, Principal Investigator, M.D., Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara Training and Research Hospital
Organization: Ankara Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraTRH-FTR-NK-09; 2023/11-090224 (Other: Ethics Committee of Traditional and Complementary Medicine, University of Health Sciences Gülhane Training and Research)
Record Dates: First submitted 2025-09-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye; Acupuncture
Keywords: Dry eye; Keratoconjunctivitis sicca; Acupuncture; Artificial tears; Ocular Surface Disease Index (OSDI); Schirmer test; Tear break-up time (tBUT); Complementary therapy
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Two-arm parallel group randomized controlled trial comparing artificial tears alone with artificial tears plus acupuncture in patients with moderate dry eye disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Tears Only (Active Comparator): Participants received topical artificial tears (sodium hyaluronate/CMC-based eye drops) according to standard treatment protocol. No additional intervention was given.
  Interventions: Drug: Artificial tears
- Experimental: Artificial Tears + Acupuncture (Experimental): Participants received artificial tears plus acupuncture therapy, administered by a certified specialist, twice weekly for 10 sessions. Each session lasted 20 minutes.
  Interventions: Drug: Artificial tears; Other: Traditional Chinese Medicine Acupuncture

INTERVENTIONS:
Drug: Artificial tears — Topical artificial tears were administered as standard therapy for moderate dry eye disease.
  Other Names: Lubricating Eye Drops; Artificial Tear Drops; Sodium Hyaluronate Eye Drops
Other: Traditional Chinese Medicine Acupuncture — Acupuncture therapy performed by a certified specialist using sterile disposable needles at predefined local and systemic acupoints (BL2, ST1, GB1, SJ23, Ex-HN5, LI4, ST36, SP6, LIV3, GB37, GB40, Ex-HN3, Du23, BL64). Sessions were delivered twice weekly for a total of 10 sessions, each lasting 20 minutes. Deqi sensation was obtained by manual stimulation. No additional systemic or topical treatments were provided to participants in this arm.
  Other Names: Needle Acupuncture; Manual Acupuncture
  Arms: Experimental: Artificial Tears + Acupuncture

SUMMARY:
This randomized clinical trial was designed to evaluate the effectiveness of acupuncture combined with artificial tears compared to artificial tears alone in patients with moderate dry eye disease. A total of 90 participants were enrolled at the University of Health Sciences, Ankara Training and Research Hospital. Patients were randomly assigned to receive either artificial tears only or artificial tears with acupuncture. Acupuncture was performed twice weekly for ten sessions by a certified specialist.

Assessments were conducted at baseline, after treatment, and at one-month follow-up using the Ocular Surface Disease Index (OSDI), Schirmer test, and tear break-up time (tBUT). The primary outcome measure was the change in OSDI score, while secondary outcomes included Schirmer test values and tBUT.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a chronic ocular surface disorder characterized by instability of the tear film, ocular discomfort, and visual disturbance. It significantly impairs quality of life, limiting daily activities such as reading, driving, and computer use. Standard treatments, including artificial tears and anti-inflammatory agents, often provide only partial or temporary relief and may not adequately address the underlying inflammatory mechanisms. As a complementary approach, acupuncture has been suggested to improve lacrimal gland function, enhance tear secretion, and reduce ocular inflammation, yet comparative evidence in moderate DED remains limited.

The aim of this study was to evaluate the short-term efficacy of acupuncture combined with artificial tears compared to artificial tears alone in patients with moderate DED. This prospective, randomized, controlled, parallel-group trial was conducted at the University of Health Sciences, Ankara Training and Research Hospital. Ninety adults aged 18-65 years, diagnosed with moderate DED according to TFOS DEWS II criteria (Schirmer 5-10 mm and tear break-up time 6-10 seconds), were enrolled between January 2024 and May 2025. Participants were randomly allocated to two groups: Group 1 received artificial tears only, while Group 2 received artificial tears plus acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of moderate dry eye disease according to TFOS DEWS II criteria
* Anesthetized Schirmer test result between 5-10 mm
* Tear break-up time (tBUT) between 6-10 seconds
* Ocular Surface Disease Index (OSDI) score ≥ 13
* Symptom duration of at least 3 months
* Signed informed consent form

Exclusion Criteria:

* Sjögren's syndrome, active blepharitis, or meibomian gland dysfunction
* Systemic rheumatologic, autoimmune, or metabolic disease (e.g., diabetes)
* Use of systemic or topical treatment for dry eye within the last 6 months
* Previous ocular surgery
* Contact lens use
* Pregnancy or lactation
* History of neurological or psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Score | Baseline (Day 1); End of Treatment (Week 5, after 10 sessions); 1-Month Follow-up (Week 9)
  The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire used to assess the severity of dry eye symptoms and their impact on visual function. Scores range from 0 to 100, with higher scores indicating more severe disease. The primary outcome is the change in OSDI score from baseline to post-treatment and 1-month follow-up.

SECONDARY OUTCOMES:
Change in Schirmer Test Values | Baseline (Day 1); End of Treatment (Week 5, after 10 sessions); 1-Month Follow-up (Week 9)
  The Schirmer test measures tear production using a standardized filter paper strip placed in the lower eyelid for 5 minutes. Values are recorded in millimeters of wetting. Lower scores indicate reduced tear secretion. The outcome is the change in tear production over time.
Change in Tear Break-Up Time (tBUT) | Baseline (Day 1); End of Treatment (Week 5, after 10 sessions); 1-Month Follow-up (Week 9)
  Tear break-up time (tBUT) is assessed after instillation of fluorescein dye. The interval between the last blink and the first appearance of a dry spot on the corneal surface is measured in seconds. Shorter times indicate instability of the tear film. The outcome is the change in tBUT values across time points.

CONTACTS AND LOCATIONS:
Overall Officials: Nadide Koca, Principal Investigator — Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital Ankara, Altindag, Turkey, 06230, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the trial was conducted as a single-center interventional study and includes sensitive clinical information that cannot be sufficiently de-identified for open sharing. Aggregate results will be reported in peer-reviewed publications.

REFERENCES:
- [Background] Duan H, Zhou Y, Ma B, Liu R, Yang T, Chu H, Huo Z, Qi H. Effect of Acupuncture Treatment on the Ocular Pain, Mental State and Ocular Surface Characteristics of Patients with Dry Eye Disease: A Non-Randomized Pilot Study. Clin Ophthalmol. 2024 Oct 3;18:2751-2764. doi: 10.2147/OPTH.S476573. eCollection 2024. PMID 39376907
- [Background] Zhang X, Zhang B, Peng S, Zhang G, Ma J, Zhu W. Effectiveness of acupuncture at acupoint BL1 (Jingming) in comparison with artificial tears for moderate to severe dry eye disease: a randomized controlled trial. Trials. 2022 Jul 27;23(1):605. doi: 10.1186/s13063-022-06486-4. PMID 35897025
- [Background] Wang Y, Peng J, Xiao L, Deng Y, Lu J, Zhou YS, Yang YJ, Peng QH. Effectiveness of acupuncture combined with artificial tears in managing dry eye syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2024 Jan 5;103(1):e36374. doi: 10.1097/MD.0000000000036374. PMID 38181299
- [Background] Moon SY, Chung HS, Lee JH, Lee H, Tchah H, Kim JY. Effectiveness of cyclosporine nanoemulsion eye drops in patients with mild-to-moderate dry eyes: objective and subjective evaluation. BMC Ophthalmol. 2024 Sep 9;24(1):401. doi: 10.1186/s12886-024-03620-5. PMID 39251947
- [Background] Bawazeer AM, Hodge WG. One-minute schirmer test with anesthesia. Cornea. 2003 May;22(4):285-7. doi: 10.1097/00003226-200305000-00001. PMID 12792467
- [Background] Kuang H, Zhu X, Chen H, Tang H, Zhao H. The immunomodulatory mechanism of acupuncture treatment for ischemic stroke: research progress, prospects, and future direction. Front Immunol. 2024 May 2;15:1319863. doi: 10.3389/fimmu.2024.1319863. eCollection 2024. PMID 38756772
- [Background] Oh JE, Kim SN. Anti-Inflammatory Effects of Acupuncture at ST36 Point: A Literature Review in Animal Studies. Front Immunol. 2022 Jan 12;12:813748. doi: 10.3389/fimmu.2021.813748. eCollection 2021. PMID 35095910
- [Background] McCann P, Kruoch Z, Lopez S, Malli S, Qureshi R, Li T. Interventions for Dry Eye: An Overview of Systematic Reviews. JAMA Ophthalmol. 2024 Jan 1;142(1):58-74. doi: 10.1001/jamaophthalmol.2023.5751. PMID 38127364
- [Background] McMonnies CW. Why the symptoms and objective signs of dry eye disease may not correlate. J Optom. 2021 Jan-Mar;14(1):3-10. doi: 10.1016/j.optom.2020.10.002. Epub 2020 Nov 23. PMID 33243674
- [Background] Villani E, Campagna G, Gentili V, Postorino EI, Genovese P, Palino P, Maini G, Carbucicchio A, Ferioli E, Nucci P, Rizzo R, Aragona P. Hydroxypropyl-Methylcellulose and GlicoPro(R) Eyedrops in the Treatment of Dry Eye Disease: In Vitro and Clinical Study. Ophthalmol Ther. 2025 Apr;14(4):787-803. doi: 10.1007/s40123-025-01101-6. Epub 2025 Mar 1. PMID 40024993
- [Background] Cartes C, Aravena C, Monsalve A, Segovia C, Romero C, Quidel D, Cid F, Monsalve R, Navarro L, Araya D, Araneda D, Sepulveda M. Prevalence of Dry Eye Disease in Laser-Assisted In Situ Keratomileusis Candidates. Eye Contact Lens. 2024 Jul 1;50(7):305-310. doi: 10.1097/ICL.0000000000001095. Epub 2024 May 2. PMID 38918902
- [Background] Chen A, Augello P, Asbell P, Ying GS; DREAM Research Group. The repeatability of tests for dry eye signs and symptoms in the dry eye assessment and management (DREAM) study. Cont Lens Anterior Eye. 2025 Apr;48(2):102322. doi: 10.1016/j.clae.2024.102322. Epub 2024 Oct 30. PMID 39477774
- [Background] Qian L, Wei W. Identified risk factors for dry eye syndrome: A systematic review and meta-analysis. PLoS One. 2022 Aug 19;17(8):e0271267. doi: 10.1371/journal.pone.0271267. eCollection 2022. PMID 35984830
- [Background] Kwon J, Moghtader A, Kang C, Bibak Bejandi Z, Shahjahan S, Alzein A, Djalilian AR. Overview of Dry Eye Disease for Primary Care Physicians. Medicina (Kaunas). 2025 Mar 6;61(3):460. doi: 10.3390/medicina61030460. PMID 40142272
- [Background] Mathebula SD, Khosa PR, Maleswene MM. Comparison of patient reported dry eye symptoms as evaluated by the ocular surface disease index and symptom assessment. Afr J Prim Health Care Fam Med. 2025 May 21;17(1):e1-e7. doi: 10.4102/phcfm.v17i1.4861. PMID 40459105
- [Background] Bhatt K, Singh S, Singh K, Kumar S, Dwivedi K. Prevalence of dry eye, its categorization (Dry Eye Workshop II), and pathological correlation: A tertiary care study. Indian J Ophthalmol. 2023 Apr;71(4):1454-1458. doi: 10.4103/IJO.IJO_2591_22. PMID 37026281
- [Background] Britten-Jones AC, Wang MTM, Samuels I, Jennings C, Stapleton F, Craig JP. Epidemiology and Risk Factors of Dry Eye Disease: Considerations for Clinical Management. Medicina (Kaunas). 2024 Sep 5;60(9):1458. doi: 10.3390/medicina60091458. PMID 39336499
- [Background] Bhujbal S, Rupenthal ID, Steven P, Agarwal P. Inflammation in Dry Eye Disease-Pathogenesis, Preclinical Animal Models, and Treatments. J Ocul Pharmacol Ther. 2024 Dec;40(10):638-658. doi: 10.1089/jop.2024.0103. Epub 2024 Oct 2. PMID 39358844
- [Background] Sheppard J, Shen Lee B, Periman LM. Dry eye disease: identification and therapeutic strategies for primary care clinicians and clinical specialists. Ann Med. 2023 Dec;55(1):241-252. doi: 10.1080/07853890.2022.2157477. PMID 36576348
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335